CLINICAL TRIAL: NCT05795426
Title: Investigation of Kinesiophobia in Volleyball Players by Gender
Brief Title: An Investigation Of Kinesiophobia in Volleyball Players, With A Focus On Gender-Based Differences
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: Volleyball Players
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Volleyball Player
Keywords: Kinesiophobia
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female volleyball players: Female volleyball players were included in the first group.
- Male volleyball players: Male volleyball players are included in the second group

SUMMARY:
Kinesiophobia is a form of behavior that includes fear and anxiety in which the person tends to stay away from the movement. . In the future, this may lead to a decrease in muscle strength and condition, leading to loss or decrease in physical adequacy, avoidance of exercise and, accordingly, psychological problems. Kinesiophobia also negatively affects the success of the treatment process in athletes or normal patients.

DETAILED DESCRIPTION:
In athletes, this situation affects the sports activity that they place at the center of their lives, causing loss of performance and, accordingly, the emergence of psychological problems. Athletes are faced with the deterioration of bone integrity during training or matches according to their branches, or they are injured by structures such as muscles, tendons and ligaments.

One of the important criteria in pain, kinesiophobia and exercise is sleep quality. Results such as sleep quality or increased stress level in insomnia and inattention may have an effect on pain or kinesiophobia. The deterioration in sleep quality leads to a decrease in the performance ability of the person, affecting the daily activity, decreasing the energy level and being in a daytime sleepy state.

ELIGIBILITY:
Inclusion criteria:

* Being between the ages of 18-30
* Taking part in Amateur Volleyball clubs

Exclusion criteria:

* Individuals under the age of 18
* Individuals who have had a surgical procedure in the last six months
* Use of NSAIDs and similar disease-modifying drugs (Diaserein, Glucosamine, etc.) in the last month.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Study Population: Amateur volleyball players will be included in the study. Individuals who will participate in the study will be reached via social media, whatsapp and message. A questionnaire will be sent to the participants via the Google search engine and they will be asked to fill it out.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale: | one day
  Tampa Kinesiophobia Scale; movement is a 17-item scale developed to measure the fear of re-injury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities.
  A 4-point Likert scoring (1=I strongly disagree, 4=I totally agree) is used in the scale. After reversing items 4, 8, 12 and 16, a total score is calculated. The person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Fatigue Severity Scale | one day
  Fatigue severity scale; It consists of 9 questions and questions the effects of one's fatigue on daily life. Each question has a score between 0 and 7. During the calculation, the arithmetic average of the total score is taken.A high score on the scale indicates a high level of fatique
Pittsburgh Sleep Quality Scale | one day
  The survey assesses the person's sleep quality over the past month. It consists of a total of 24 questions, 19 of which are filled in by the person filling out the questionnaire, and 5 of them are filled by the participant's roommate or bed partner if they have a bed partner. While calculating the index, the questions answered by the spouse and friend of the person are not included in the calculation. In the scoring of the index; There are 7 components: subjective sleep quality, sleep latency (latency), sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. A high score on the scale indicates a high level of slepp problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçeşehir University, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)

REFERENCES:
- [Background] Watanabe K, Koshino Y, Kawahara D, Akimoto M, Mishina M, Nakagawa K, Ishida T, Kasahara S, Samukawa M, Tohyama H. Kinesiophobia, self-reported ankle function, and sex are associated with perceived ankle instability in college club sports athletes with chronic ankle instability. Phys Ther Sport. 2023 May;61:45-50. doi: 10.1016/j.ptsp.2023.02.008. Epub 2023 Feb 26. PMID 36871492